CLINICAL TRIAL: NCT00158561
Title: An Open-label Three Arm Trial of the Efficacy and Safety of Chlorproguanil / Dapsone (Lapdap) Compared With Chloroquine and Sulfadoxine / Pyrimethamine for the Treatment of Vivax Malaria in Pakistan and Afghanistan
Brief Title: Chlorproguanil/Dapsone Compared With Chloroquine and SP for Vivax Malaria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: HealthNet TPO (Other)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: ITDCKD45
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Malaria; Vivax Malaria
Keywords: vivax; treatment; Asia
MeSH Terms: conditions — Malaria; Malaria, Vivax | interventions — fanasil, pyrimethamine drug combination; chloroguanil, dapsone drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: sulfadoxine-pyrimethamine and chlorproguanil-dapsone

SUMMARY:
To determine whether two cheap antifolates (chlorproguanil-dapsone and sulfadoxine-pyrimethamine) which work against falciparum malaria in this region are sufficiently effective against vivax malaria to be deployed in areas where diagnosis is poor and the burden of malaria is high, a randomised controlled trial of the three drugs is being undertaken comparing their efficacy in treating malaria.

DETAILED DESCRIPTION:
Objectives:

Primary:

To evaluate the comparative efficacy of chlorproguanil / dapsone with sulfadoxine-pyrimethamine for the treatment of vivax malaria in Pakistan and eastern Afghanistan.

Secondary:

* To compare the efficacy of chlorproguanil-dapsone and sulfadoxine-pyrimethamine with chloroquine
* To evaluate the safety profile of chlorproguanil / dapsone in south Asians from this region when used for the treatment of vivax malaria.
* To evaluate the effect of chlorproguanil / dapsone on gametocyte clearance rates.
* To evaluate the effect of chlorproguanil / dapsone on subsequent relapse due to vivax malaria.

Study Population:

750 P.vivax positive individuals recruited from the Malaria Reference Centre in Jalalabad, Afghanistan and at health facilities in Afghan refugee camps in North West Frontier Province (NWFP), Pakistan supervised by HealthNet International

Efficacy Parameters :

Primary Efficacy Variable:

• Day 14 slide clearance rate (complete clearance of parasites), assessed by microscopists who are blind to treatment allocation. Slides will be double read.

Secondary Efficacy Variables

* Day 28 slide clearance rate defined as the number of treated patients with clearance of parasitaemia within 14 days of starting treatment, without subsequent recrudescence up to day 28.
* Day 14 clinical failure rate (presence of symptoms of malaria in the presence of parasitaemia).
* Day 28 clinical failure rate.
* Adverse events.
* Haemoglobin level increased by at least 1g/dl by day 14.
* Clearance of gametocytaemia by day 3, 7, and 14.
* Number of subsequent malaria episodes in next 6 months. It is assumed that the population of each treatment arm is equally likely to be re-infected in this time scale. Therefore any measurable difference in number of subsequent episodes between treatment arms will be due to a relapse.
* In G6PD deficient patients the change in mean haemoglobin.

Safety Parameters:

Adverse events and laboratory findings will be monitored in all patients. Regular haemoglobin to identify haemolysis.

Study design:

Recruitment and administration:

Recruitment and administration of all treatments will be directly observed by the trial coordinator and trial pharmacist, and/or health unit clinician.

Dosing Schedules:

Chlorproguanil-dapsone (Lapdap): (target doses 2.0 and 2.5 mg/kg respectively) daily for 3 days .

Sulfadoxine - pyrimethamine (SP): (target doses 1.25 and 25.0 mg/kg respectively) once only.

Chloroquine (CQ): (target dose 25mg/kg ) daily for 3 days.

Follow up:

Patients will return to the clinic on days 0, 1, 2, 3, 7, 14, 21 and 28 for supervised dosing, thick and thin smears, blood spot filter papers, update of clinical record forms, determination of haemoglobin, full blood cell counts, liver function tests, determination of adverse events and concomitant medication details, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Presentation at BHU or clinic with probable clinical malaria.
2. Infection with P. vivax, confirmed by microscopy.
3. Age 3 years or older (no restriction on upper age limit).
4. Written or witnessed verbal consent obtained from the patient or the patients parent or guardian.
5. Married women of child bearing age confirmed to be non-pregnant at outset and willing to remain thus for the duration of the study.
6. Willingness to comply with the requirements of the protocol and particularly to provide venous and thumb prick blood samples.
7. Available for follow up for the duration of the study and not less than 6 months.
8. Willingness to report to the BHU or clinic if they feel unwell in the 6 months following completion (i.e. 7 months from enrolment date). NB these patients will only be those recruited up to 7 months before the end of the study period.
9. Availability of G6PD status by willingness to be tested at admission.

Exclusion Criteria:

1. General condition requiring hospital admission.
2. Evidence of any concomitant infection likely to mask treatment response at the time of presentation.
3. Presence of any other underlying disease that compromises the diagnosis and the evaluation of the response to the study medication.
4. History of allergy to sulphonamides, dapsone or chloroquine or hypersensitivity to biguanides (eg proguanil, chlorproguanil) sulphones (eg frusemide, thiazides, acetazolamide, and sulphonylureas) or any other tablet contents.
5. Known methaemoglobin reductase deficiency and haemoglobin M.
6. Treatment within the past twenty-eight days with sulfadoxine/pyrimethamine (Fansidar), sulfalene/pyrimethamine (Metakelfin), mefloquine-sulfadoxine-pyrimethamine (Fansimef); 21-days with mefloquine, or 7-days with amodiaquine, chloroquine, halofantrine, quinine (full course), primaquine, atovaquone - proguanil, artemisinin derivatives, co-artemether, trimethoprim, chloramphenicol, erythromycin, tetracycline or clindamycin.
7. Visible jaundice.
8. Use of an investigational drug within 30 days or 5 half-lives whichever is the longer.
9. Severe anaemia (Hb<7 g/dl).
10. Other species of malaria seen.
11. Pregnancy, assessed by pregnancy test in all married women of child-bearing age (age over 14 and under 50).

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 750
Dates: Start 2004-02; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Day 14 slide clearance rate (complete clearance of parasites), assessed by microscopists who are blind to treatment allocation.

SECONDARY OUTCOMES:
Day 28 slide clearance rate defined as the number of treated patients with clearance of parasitaemia within 14 days of starting treatment, without subsequent recrudescence up to day 28.
Day 14 clinical failure rate (presence of symptoms of malaria in the presence of parasitaemia).
Day 28 clinical failure rate.
Adverse events.
Haemoglobin level increased by at least 1g/dl by day 14.
Clearance of gametocytaemia by day 3, 7, and 14.
Number of subsequent malaria episodes in next 6 months. It is assumed that the population of each treatment arm is equally likely to be re-infected in this time scale. Therefore any measurable difference in number of subsequent episodes between treatment
In G6PD deficient patients the change in mean haemoglobin.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Whitty, FRCP, Principal Investigator — London School of Hygiene and Tropical Medicine; Mark Rowland, PhD, Study Director — London School of Hygiene and Tropical Medicine
Locations (1):
- HealthNet International, Peshawar, Pakistan

REFERENCES:
- [Result] Leslie T, Mayan MI, Hasan MA, Safi MH, Klinkenberg E, Whitty CJ, Rowland M. Sulfadoxine-pyrimethamine, chlorproguanil-dapsone, or chloroquine for the treatment of Plasmodium vivax malaria in Afghanistan and Pakistan: a randomized controlled trial. JAMA. 2007 May 23;297(20):2201-9. doi: 10.1001/jama.297.20.2201. PMID 17519409